

# Statistical Analysis Plan

| Protocol Number/version | DBC-18PENDL02/Version 4.0 25Feb2019 |
|---|---|
| Protocol Title | Comparative User Experiences with BD Nano <sup>™</sup> PRO 4mm × 32G Extra |
| | Thin Wall Pen Needle vs the Artsana Insupen <sup>®</sup> Extr3me $4\text{mm} \times 33\text{G}$ , Art- |
| | sana Insupen $^{\circledR}$ Extr3me 3.5mm $	imes$ 34G and the Simple Diagnostics Comfort |
| | $\mathrm{EZ}^{\scriptscriptstyleTM}$ 4mm $	imes$ 33G Pen Needles |
| SAP Date | May 30, 2019 |
| Version History | March 5, 2019: Original Release |
| | May 14, 2019: Additional analysis for site effect was added in Section 6.2.1 to |
| | 6.2.4. Potential DBC-18PENDL01 and DBC-18PENDL02 combined analy- |
| | sis was added in Section 6.2.1.1, 6.2.2.1, 6.2.3.1 and 6.2.4. |

This document is proprietary to Becton Dickinson. No part of it may be distributed or shared with persons other than BD associates without written permission from Global Clinical Development (GCD).

# Approval

| Signature below indicates appro- | Signature below indicates approval of the statistical analysis plan as written. | |
|---|---|---|
| Function | Name | Signature |
| Study Statistician (Author) | Wen Yue | This document is signed electronically in the eTMF system. |
| Associate Director, Statistics | Julie Bérubé | This document is signed electronically in the eTMF system. |
| Medical Affairs Team | Shahista Whooley | This document is signed electronically |
| Representative | | in the eTMF system. |
| Study Manager | Lydia Blank | This document is signed electronically in the eTMF system. |

DBC-18PENDL02 



# Contents

| O | | tudy Description |
|---|---|---|
| 2. | | Background |
| 2. | • | Objectives |
| 2. | _ | Design |
| 2. | _ | oints |
| | 2.4.1 | Primary Endpoints |
| | 2.4.2 | Secondary Endpoints |
| | 2.4.3 | Exploratory Endpoints |
| | 2.4.4 | Safety Endpoints |
| 2. | _ | otance Criteria |
| | 2.5.1 | Primary Objective |
| | 2.5.2 | Secondary Objectives |
| | 2.5.3 | Exploratory Objectives |
| $\mathbf{S}$ | ample S | ize |
| Iı | ntended | Statistical Software |
| Ъ | ata | |
| ப | ala | |
| | 1 Dotok | agga Information |
| 5. | | pase Information |
| | | pase Information |
| 5.<br>5. | 2 Analy tatistica | rsis Population Set(s) |
| 5.<br>5. | 2 Analy tatistica 1 Derive | rsis Population Set(s) |
| 5.<br>5. | 2 Analy tatistical 1 Derive 6.1.1 | rsis Population Set(s) |
| 5.<br>5.<br><b>S</b> | 2 Analy tatistica 1 Derive 6.1.1 6.1.2 | Sis Population Set(s) |
| 5.<br>5.<br><b>S</b> ·<br>6. | 2 Analy tatistica 1 Derive 6.1.1 6.1.2 6.1.3 | rsis Population Set(s) |
| 5.<br>5. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy | rsis Population Set(s) I Analysis / Calculations ed Variables |
| 5.<br>5.<br><b>S</b><br>6. | 2 Analy tatistica 1 Derive 6.1.1 6.1.2 6.1.3 | Sis Population Set(s) I Analysis / Calculations ed Variables Relative VAS Scale Leakage Scale Injection force Sis Method Analysis of Injection pain |
| 5.<br>5.<br><b>S</b> ·<br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy 6.2.1 | Sis Population Set(s) I Analysis / Calculations ed Variables |
| 5.<br>5.<br><b>S</b> ·<br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy | Relative VAS Scale Leakage Scale Injection force sis Method Analysis of Injection pain 6.2.1.1 Additional analysis Analysis of Injection force |
| 5.<br>5.<br><b>S</b><br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy 6.2.1 6.2.2 | Sis Population Set(s) I Analysis / Calculations ed Variables |
| 5.<br>5.<br><b>S</b><br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy 6.2.1 | I Analysis / Calculations ed Variables Relative VAS Scale Leakage Scale Injection force sis Method Analysis of Injection pain 6.2.1.1 Additional analysis Analysis of Injection force 6.2.2.1 Additional analysis Analysis of Needle Bending and Leakage |
| 5.<br>5.<br><b>S</b><br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy 6.2.1 6.2.2 6.2.3 | I Analysis / Calculations ed Variables |
| 5.<br>5.<br><b>S</b><br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy 6.2.1 6.2.2 | Relative VAS Scale |
| 5.<br>5.<br><b>S</b><br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy 6.2.1 6.2.2 6.2.3 | I Analysis / Calculations ed Variables |
| 5.<br>5.<br><b>S</b><br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy 6.2.1 6.2.2 6.2.3 | I Analysis / Calculations ed Variables |
| 5.<br>5.<br><b>S</b> ·<br>6. | 2 Analy tatistical 1 Derive 6.1.1 6.1.2 6.1.3 2 Analy 6.2.1 6.2.2 6.2.3 | I Analysis / Calculations ed Variables |

DBC-18PENDL02 



| 8 | Exa | mple i | Reports | 14 |
|---|------------|--------|-------------------------------|----|
| | 8.1 | Study | Execution | 15 |
| | | 8.1.1 | Analysis Population Set(s) | 15 |
| | | 8.1.2 | Data Exclusions | 15 |
| | | 8.1.3 | Executive Summary | 16 |
| | 8.2 | Analy | rsis and Results | 17 |
| | | 8.2.1 | Injection Pain | 17 |
| | | 8.2.2 | Injection force | 19 |
| | | 8.2.3 | Needle Bending | 21 |
| | | 8.2.4 | Leakage from Injection Site | 21 |
| | | 8.2.5 | Exploratory Objectives | 23 |
| | 8.3 | Demo | graphics and Diabetes History | 23 |
| 9 | App | oendix | | 25 |
| | $9.1^{-1}$ | Discor | ntinued Data | 25 |
| | 9.2 | | ng Data | 25 |
| | 9.3 | | ese Events | 25 |

DBC-18PENDL02 



# 1 List of Abbreviations and Definitions

- **AE:** Adverse event
- **BD:** Becton Dickinson and Company
- GCD: Global Clinical Development, BD
- CI: Confidence Interval
- CRF: Case Report/Record Form
- **G**: Gauge
- **IFU:** Instruction for Use
- NI: Non Inferiority
- VAS: Visual Analog Scale
- RS: Randomization schedule
- SAE: Serious Adverse Event
- SAP: Statistical Analysis Plan
- **SD:** Standard Deviation

DBC-18PENDL02 



# 2 Overall Study Description

### 2.1 Study Background

Pen needles are a component of pen-based injection systems routinely utilized for parenteral administration of medications such as insulin. In 2010, BD introduced a 4mm  $\times$  32G pen needle. At that time it was the shortest and thinnest pen needle available. In addition to lowering the risk for intramuscular injections, this pen needle was demonstrated to be preferred by patients vs. their current pen needles. Since its introduction, competitors have launched similar length pen needles with thinner gauge needles, such as 33G and 34G. The intent of this comparative use study is to determine whether patient experiences are different when using the BD Nano<sup>TM</sup> PRO 4mm  $\times$  32G extra thin wall, 5-bevel pen needle (herein referred to as BD Nano<sup>TM</sup> PRO) vs competitive thinner pen needles - Artsana Insupen<sup>®</sup> Extr3me 4mm  $\times$  33G, Artsana Insupen<sup>®</sup> Extr3me 3.5mm  $\times$  34G and the Simple Diagnostics Comfort EZ<sup>TM</sup> 4mm  $\times$  33G Pen Needles (herein referred to as comparators). These experiences include injection pain, force to deliver dose, bending, and ability to deliver full dose (leakage).

# 2.2 Study Objectives

#### • Primary Objective

Demonstrate non-inferiority of the BD Nano<sup>TM</sup> PRO pen needle compared to each of three (3) commercially available comparators (33G and 34G) for injection pain.

#### • Secondary Objectives

Demonstrate superiority of BD Nano<sup>™</sup> PRO vs each of 3 comparator pen needles for the following:

- 1. Leakage from the needle tip and the injection site (measurements combined) after removal from body
- 2. Subject perceived force required to deliver dose
- 3. Patient end needle bending after removal from body
- 4. If primary outcome demonstrates non-inferiority then evaluate for superiority of BD Nano<sup>™</sup> PRO vs each comparator.

#### • Exploratory Objectives

Compare BD Nano<sup>™</sup> PRO vs each of 3 comparator pen needles for the following:

- 1. Injection time
- 2. Patient end needle breaking at any time
- 3. Survey responses pertaining to subjective assessments of pen needle characteristics

DBC-18PENDL02 



# 2.3 Study Design

This is a subject partially blinded, block randomized, prospective, single-visit, multi-center study to compare user experiences with BD Nano™ PRO pen needle vs. three (3) thinner commercially available comparator pen needles (Artsana Insupen® Extr3me 33G, Artsana Insupen® Extr3me 34G and the Simple Diagnostics Comfort EZ™ 33G Pen Needles). The study will include up to 146 study subjects having Type 1 or Type 2 diabetes. Study conduct will consist of one 60 to 120 minute site visit in which pre-set doses of saline will be abdominally delivered by subjects via a reusable insulin pen device. All pen needles will be attached by study staff and pen needle outer cover and inner shield will be removed for subjects. Subjects are to perform 12 injections into the abdomen (6 pairs of injections). Pairs of injections will be evaluated and each pair will contain one BD Nano™ PRO and one comparator pen needle. Within the 12 injections, each comparator will be injected twice, therefore each subject will experience 2 of each of the following pairs:

- ullet BD Nano PRO pen needle vs Artsana Insupen Extr3me 4mm  $\times$  33G  $\times$  2
- $\bullet$ BD Nano  $^{\mathbb{M}}$ PRO pen needle v<br/>s Artsana Insupen ® Extr3me 3.5mm × 34G × 2
- BD Nano<sup>TM</sup> PRO pen needle vs Simple Diagnostics Comfort  $\mathrm{EZ}^{\mathrm{TM}}$  4mm  $\times$  33G  $\times$  2

Subjects will not see pen needle labels or be informed which pen needle is being used to inject. The BD Nano™ PRO has a distinct configuration and subjects will most likely notice the difference vs the comparators. Subjects will not be informed of the BD's or the comparator's pen needle brand, length or gauge. The pen needle order within the pairs of injections will be randomized for each subject and the pairs will be randomized to various abdominal injection sites within each subject. Besides being informed of the requirement to insert the pen needles "straight-in" (perpendicular), subjects will be instructed to use their usual injection technique.

#### 2.4 Endpoints

## 2.4.1 Primary Endpoints

**Injection Pain**: Each Subject will evaluate pain after completion of each pair of injections using a 15 cm relative Visual Analog Scale (VAS).

#### 2.4.2 Secondary Endpoints

After each injection:

- Leakage: After saline delivery equivalent to 30U of U100 insulin (0.3mL) and subject removal of pen needle from body, study staff will use the provided materials and scale to absorb leakage from the pen needle tip and injection site to measure the amount of leakage.

  Leakage will be considered to be present if measurement is equivalent to or greater than 5% of dose (equivalent to ≥ 0.015q).
- Needle bending: Study staff will use a provided needle bend scale and visually inspect retained pen needles to determine the presence of bending. If present, study staff will determine and document degree of bend with the provided scale. For the purpose of answering the study objective, needle bend will be considered if the bend rating > 2.

DBC-18PENDL02 



#### After each pair of injections:

• Injection force: Each subject will evaluate perceived injection force after each pair of injections using a 5-point Likert scale (from 1st injection required much less force to deliver medication to 2nd injection required much less force to deliver medication).

#### 2.4.3 Exploratory Endpoints

During each injection: Injection time - includes the following time periods for each injection

- Time from when subject first pushes injection button to time button fully depressed (delivery time)
- Time from when injection button fully depressed to when pen needle removed from body
- Total injection time the 2 time periods above combined

#### After each injection:

• Breaking: Study Staff will record any patient end needle breakage. Breakage is defined as the patient-end metal cannula separated into two pieces.

#### After all injections completed:

- Survey responses: Subject completes a 5-point Likert scale survey (from Disagree to Agree). Subject will be instructed to respond to the questions based on their usual (in-home use) injection experience. Subject responses to survey questions will be tallied. The survey includes the following four questions:
  - 1. Injection pain affects my level of satisfaction with my treatment.
  - 2. Injection pressure needed to deliver the dose affects my level of satisfaction with my treatment.
  - 3. Post injection leakage increases my level of concern that I may not be receiving my full dose of medication.
  - 4. A bent needle increases my level of concern about the reliability of my injection.

#### 2.4.4 Safety Endpoints

Occurrence of adverse events will be evaluated, recorded, and followed up as required.

### 2.5 Acceptance Criteria

#### 2.5.1 Primary Objective

BD Nano<sup>TM</sup> PRO non-inferior to each comparator for injection pain with partially blinded injections based on relative VAS, where -75mm indicates worse pain for BD Nano<sup>TM</sup> PRO and +75mm indicates worse pain for comparator with a non-inferiority criterion of -10mm.

DBC-18PENDL02 



#### 2.5.2 Secondary Objectives

- The BD Nano<sup>™</sup> PRO will be evaluated for superiority vs each comparator for leakage, injection force, and bending.
- If the BD Nano<sup>™</sup> PRO demonstrates non-inferiority for injection pain for the Primary Objective, compare the BD Nano<sup>™</sup> PRO vs each comparator for superiority.

#### 2.5.3 Exploratory Objectives

No formal acceptance criterion has been established for the following objectives - time to deliver dose, total injection time, and survey responses after all injections completed.

# 3 Sample Size

Pain: Assuming the SD for relative VAS is around 50mm (based on DBC-17NUCLS07), a sample size of 266 pairs per each comparator has >90% power of passing a -10mm NI criteria, assuming no true difference in pain (based on a 2-sided 95% CI for the mean).

Leakage: Based on previous study data (BDT-2P00116) where leakage was greater than or equal to 1.5U was observed in 66/298 (22.1%) of injections performed with Artsana 34G, in 25/299 (8.4%) of injections performed with Comfort EZ 33G, in 19/296 (6.4%) of injections performed with Artsana 33G and in 3/297 (1%) of injections performed with BD Nano™ PRO, a simulation was performed (code found in SVN repository under DBC-18PENDL01/Sample Size/Bayesian prior proportion.R) indicating that 798 injections with BD Nano™ PRO and 266 injections per each comparator would provide >90% power to show BD Nano™ PRO superiority to each comparator. So the number of subjects needed is 133.

A 10% buffer was added (to compensate for subject attrition or unusable data), leading to a planned enrollment number of 146 subjects.

#### 4 Intended Statistical Software

This document was generated with R version 3.5.1 (2018-07-02) and the following packages (version) were used: assertthat (0.2.0), base (3.5.1), BDbasics (0.2.4), bindr (0.1.1), bindrcpp (0.2.2), colorspace (1.3.2), compiler (3.5.1), crayon (1.3.4), datasets (3.5.1), dplyr (0.7.6), ggplot2 (3.1.1), glue (1.3.0), graphics (3.5.1), grDevices (3.5.1), grid (3.5.1), gtable (0.2.0), lattice (0.20.35), lazyeval (0.2.1), magrittr (1.5), methods (3.5.1), munsell (0.5.0), nlme (3.1.137), pillar (1.3.0), pkgconfig (2.0.2), plyr (1.8.4), purrr (0.2.5), R6 (2.2.2), Rcpp (0.12.18), reshape2 (1.4.3), rJava (0.9.10), rlang (0.2.2), scales (1.0.0), stats (3.5.1), stringi (1.1.7), stringr (1.3.1), tibble (1.4.2), tidyselect (0.2.4), tools (3.5.1), utils (3.5.1), withr (2.1.2), xlsx (0.6.1), xlsxjars (0.6.1), xtable (1.8.3).

The analysis of this study will be conducted within the same environment or using more recent versions.

DBC-18PENDL02 



### 5 Data

#### 5.1 Database Information

The input data will consist in several csv (comma separated values) files exported from Clindex.

Files will be saved in

https://svn.bdx.com:8443/svn/stats\_and\_dm/DM and Stats Outputs/DBC/DBC-18PENDL02/Data and read directly into R for analysis.

# 5.2 Analysis Population Set(s)

All data collected will be analyzed and reviewed for possible exclusion based on significant outliers or protocol deviations.

Injections where bleeding was observed will not be used in the leakage analyses.

Analyses of relative data will only include pairs where both injections were completed.

Demographic information and Diabetes history collected for all subjects randomized will be tabulated.

Data from all subjects will be included in the summary of safety parameters.

# 6 Statistical Analysis / Calculations

#### 6.1 Derived Variables

#### 6.1.1 Relative VAS Scale

After completion of each pair of injection, subjects will be asked to compare pain between the pen needles using a 150mm relative VAS Scale. Marks made on the 150mm relative VAS Scale are read using a 0 - 20 grid and the resulting discrete scores entered into the database. The results will be transformed to a [-75mm, 75mm] scale for analysis and reporting, where positive scores will reflect less pain for BD Nano Pro and negative scores will reflect less pain for comparator pen needle.

Subjects will draw a vertical line on a relative VAS scale for each pair of injections, to indicate their relative pain perception for the pen needle used first or second in the pair. A vertical line drawn to the left of the center mark indicates that the 1st injection was less painful. A vertical line drawn to the right of the center mark indicates that the 2nd injection was less painful. A vertical line drawn at the center mark indicates no difference. Figure 1 shows an example of a 150mm (may not be to scale) relative VAS scale.

DBC-18PENDL02 



Which injection was less painful?



Figure 1: VAS Scale for Injection Pain

The scores are entered into the database on a discrete 0-20 scale. These scores will be transformed to a 150mm VAS on a [-75mm, 75mm] scale as follows:

Let  $Y_{recorded}$  (= 0, 1,  $\cdots$ , 20) be the recorded VAS score, the first transformation for the analysis of VAS score,  $Y_{analysis}^*$  (mm), will be calculated as:

$$Y_{analysis}^* = \frac{150}{20} * Y_{recorded} - 75 \tag{1}$$

The sign of the VAS responses  $Y_{analysis}^*$  will then be adjusted depending on which pen needle was used in the first and in the second injection, so that positive scores (+) will reflect less pain for BD Nano and negative scores (-) will reflect less pain for comparator pen needles. Let  $Y_{analysis}$  be the final relative VAS score used for the analysis. Then:

$$Y_{analysis} = \begin{cases} Y_{analysis}^*, & \text{if BD Nano is provided in the 2}^{\text{nd}} & \text{injection} \\ -Y_{analysis}^*, & \text{if BD Nano is provided in the 1}^{\text{st}} & \text{injection} \end{cases}$$
(2)

#### 6.1.2 Leakage Scale

Study Staff will use the provided materials and scale to absorb leakage from the pen needle tip and injection site to measure the amount of leakage. Leakage will be considered to be present if measurement is equivalent to or greater than 5% of dose (equivalent to equal to or greater than 1.5U of U100 insulin (or 0.015g)). A binary leakage variable will be created with the equation below:

$$Y_{Leakage} = \begin{cases} \text{Yes, if recorded leakage} \ge 0.015g\\ \text{No, if recorded leakage} < 0.015g \end{cases}$$
(3)

DBC-18PENDL02 



#### 6.1.3 Injection force

Injection force will be evaluated after each pair of injections using a 5-point Likert scale and the results will be converted to ratings of -2 to 2 as below:

$$Y_{Injectionforce}^* = \begin{cases} -2, & \text{if 1st injection significantly less thumb force} \\ -1, & \text{if 1st injection slightly less thumb force} \\ 0, & \text{if no difference} \\ 1, & \text{if 2nd injection slightly less thumb force} \end{cases} \tag{4}$$

The sign of the injection force responses  $Y_{Injectionforce}^*$  will then be adjusted depending on which pen needle was used in the first and in the second injection, so that positive scores (+) will reflect less thumb force for BD Nano and negative scores (-) will reflect less thumb force for comparator pen needles. Let  $Y_{Injectionforce}$  be the final injection force score used for the analysis. Then:

$$Y_{Injectionforce} = \begin{cases} Y_{Injectionforce}^{*}, & \text{if BD Nano is provided in the 2}^{\text{nd}} & \text{injection} \\ -Y_{Injectionforce}^{*}, & \text{if BD Nano is provided in the 1}^{\text{st}} & \text{injection} \end{cases}$$
(5)

The responses will also be converted to 3 categories: favoring comparator pen needle (negative ratings), no difference (0 ratings) and favoring BD Nano™ PRO (positive ratings) with the equation below:

$$Y_{Injection force(categorical)} = \begin{cases} \text{Comparator pen needle with less injection force if recorded rating} < 0 \\ \text{No difference, if recorded rating} = 0 \\ \text{BD Nano with less injection force if recorded rating} > 0 \end{cases}$$
 (6)

DBC-18PENDL02 



### 6.2 Analysis Method

This section provides a detailed description of the statistical analysis that will be performed in this study.

Unless otherwise stated, all the statistical tests are two-sided at a significance level of 5%.

Summary statistics (number of observations, mean, 95% CI for mean, median, standard deviation and range) for all quantitative responses will be presented in tables. Frequency tables with number of observations, percentage of total will be created for all discrete responses. If a modeling approach is applied, the fitted mean with 95% CI will be presented in tables.

Bar plots may be provided for some responses.

#### 6.2.1 Analysis of Injection pain

For each comparator PN, a two-sided 95% confidence intervals will be calculated for the average rating. A modeling approach including data from all pairs of injections (all comparator PN included) will be used to analyze the data and estimate average ratings for each comparator PN adjusting for the pair order effect, BD order effect within pair (due to the often-observed bias towards favoring the last pen needle used in a pair), abdomen site effect, comparator PN effect and random subject effect. The interaction of PN and clinical site will be verified. If the interaction is significant, multiple comparisons for site difference by each PN will be conducted and results will be presented by site for PNs with significant site difference. If the interaction is not significant, it will be dropped from the model and clinical site will be included as main effect. If the site difference is significant, results will be presented by site for each PN. Otherwise, the site effect will be dropped from the model. Results will be tested for non-inferiority, followed by superiority:

- If the lower bound of the CI is > -10mm, we can conclude in non-inferiority.
- If the lower bound of the CI is > 0mm, we can conclude in superiority.

```
> ## Example for estimated pen needle subgroup means (Site effect not significant)
> ## if the lower CL is > -10, non-inferiority is satisfied
> ## if the lower CL is > 0, superiority is satisfied
> library(emmeans)
> emmeans(model.fit, ~Comparator)
```

DBC-18PENDL02 



 Comparator
 emmean
 SE
 df
 lower.CL
 upper.CL

 Artsana 33G
 26.87836
 5.747502
 140.26
 15.515420
 38.24129

 Artsana 34G
 20.09732
 7.841233
 139.57
 4.594362
 35.60027

 Simple Diagnostics
 22.40372
 6.075449
 140.25
 10.392416
 34.41502

Degrees-of-freedom method: kenward-roger

Confidence level used: 0.95

#### 6.2.1.1 Additional analysis

Given that there is no significant site effect and no significant difference between any comparator PNs, data from DBC-18PENDL02 and DBC-18PENDL01 will be combined for analysis. An overall result combining all comparators in the two studies will be presented.

#### 6.2.2 Analysis of Injection force

For each comparator PN, the responses in 5-point Likert scale will be converted to ratings of -2 to 2 (where positive ratings favor BD, see Section 6.1.3) and a two-sided 95% confidence interval will be calculated for the average rating. A modeling approach including data from all pairs of injections (all comparator PN included) will be used to analyze the data and estimate average ratings for each comparator PN adjusting for the pair order effect, BD order effect within pair (due to the often-observed bias towards favoring the last pen needle used in a pair), abdomen site effect, comparator PN effect and random subject effect. The interaction of PN and clinical site will be verified If the interaction is significant, multiple comparisons for site difference by each PN will be conducted and results will be presented by site for PNs with significant site difference. If the interaction is not significant, it will be dropped from the model and clinical site will be included as main effect. If the site difference is significant, results will be presented by site for each PN. Otherwise, the site effect will be dropped from the model.

If the lower bound of the CI for the average rating is > 0mm, we can conclude in superiority.

Responses will also be converted to 3 categories: favoring comparator pen needle (negative ratings), no difference (0 ratings) and favoring BD Nano™PRO (positive ratings) (see Section 6.1.3). The difference in percentage of responses with a preference for BD Nano vs each comparator pen needle will be calculated by Bayesian approach, adjusting for the "no preference" category.

#### 6.2.2.1 Additional analysis

Given that there is no significant site effect and no significant difference between any comparator PNs, data from DBC-18PENDL02 and DBC-18PENDL01 will be combined for analysis. An overall result combining all comparators in the two studies will be presented.

# 6.2.3 Analysis of Needle Bending and Leakage

If there is a sufficient number of occurrences for a modeling approach, analysis will be performed using a binary logistic regression with random subject effect and fixed pen needle type effect, pair order effect,

DBC-18PENDL02 



PN order effect within pair and abdomen site effect. The interaction of PN and clinical site will be verified. If the interaction is significant, multiple comparisons for site difference by each PN will be conducted and results will be presented by site for PNs with significant site difference. If the interaction is not significant, it will be dropped from the model and clinical site will be included as main effect. If the site difference is significant, results will be presented by site for each PN. Otherwise, the site effect will be dropped from the model. The average difference in percentage of occurrence with BD PN and each comparator pen needle will be calculated with 95% confidence interval and assessed for statistical significance. The upper bound of the confidence interval will be compared to 0: superiority will be concluded given that the upper bound of the 95% confidence interval for the difference in proportions is < 0%.

If a modeling approach cannot be applied, a proportion test will be used to detect the difference in percentage of occurrence between sites for each PN. If there is no significant difference, the difference in percentage of occurrence with BD PN and each comparator pen needle will be calculated with 95% confidence interval (Score method) and assessed for statistical significance.

```
PN emmean SE df asymp.LCL asymp.UCL BD Nano 0.07942998 13925529 Inf -27293535 27293535 Artsana 33G 0.07942595 8632818 Inf -16920013 16920013 Artsana 34G 0.07944491 11568566 Inf -22673973 22673973 Simple Diagnostics 0.07940803 12153341 Inf -23820110 23820111
```

Results are given on the logit (not the response) scale. Confidence level used: 0.95

#### 6.2.3.1 Additional analysis

Given that there is no significant site effect for DBC-18PENDL02, no significant difference for BD PN between DBC-18PENDL02 and DBC-18PENDL01, and no significant difference between any comparator PNs, data from DBC-18PENDL02 and DBC-18PENDL01 will be combined for analysis. An overall result combining all PNs in the two studies will be presented.

DBC-18PENDL02 



# 6.2.4 Analysis of Exploratory Objectives (Delivery time, Total injection time, Needle Breaking, and Non-Comparative Questionnaire)

### 6.2.4.1 Delivery time and Total injection time

A mixed effect model will be used (fixed effects of pen needle type, abdomen site, order of pair, order of pen needle within pair and random subject effect) to estimate average difference (BD Nano PN - each comparator PN) in delivery time and total injection time. The interaction of PN and clinical site will be verified. If the interaction is significant, comparison results will be presented by site. If the interaction is not significant, it will be dropped from the model and clinical site will be included as main effect. If the site difference is significant, mean delivery time and mean total injection time will be presented by site for each PN. Otherwise, the site effect will be dropped from the model. A Box-Cox transformation might be used to normalize the data if necessary. The upper bound of the confidence interval will be compared to 0: superiority will be concluded given that the upper bound of the 95% interval for the average difference is < 0 seconds.

Given that there is no significant site effect for DBC-18PENDL02, no significant difference for BD PN between DBC-18PENDL02 and DBC-18PENDL01, and no significant difference between any comparator PNs, data from DBC-18PENDL02 and DBC-18PENDL01 will be combined for analysis. An overall result combining all PNs in the two studies will be presented.

#### 6.2.4.2 Needle Breaking

The number and proportion of needle breaking occurrence for each pen needle type will be summarized. In addition, a 95% confidence interval for difference in proportions between BD Nano PN and each comparator PN will be calculated using the score method for independent proportions. Site effect will be verified in a similar way with needle bending.

#### 6.2.4.3 Non-Comparative Questionnaire

All the responses from Non-Comparative Questionnaire will be summarized with number and percentage of each option. Data from DBC-18PENDL02 and DBC-18PENDL01 will be combined for analysis if possible.

# 7 Safety Analysis

Data listings will be provided for any adverse events and serious adverse events in Appendix. The events will also be summarized descriptively per pen needle type. No safety analysis is planned.

# 8 Example Reports

This section provide examples of tables and graphical representations that will be provided in the study statistical report. These table examples were generated using the sample data available from the data base test framework which do not provide an exhaustive or representative example of the values and levels that will be obtained in the study. They are intended to provide illustrative examples of the tables and figures that will be included in the final statistical analysis report.

DBC-18PENDL02 



# 8.1 Study Execution

The number of subjects enrolled, randomized, withdrawn, who completed and who are excluded will be provided as in Table 2. More details on specific data may be provided in Summary Statistics and Appendix.

# 8.1.1 Analysis Population Set(s)

Table 1: Population Disposition (Example only)

| Subject.Population | N | Comments |
|----------------------------------------|-----|--------------|
| Subjects Enrolled | 252 | none |
| Subjects who did not meet I/E Criteria | 6 | none |
| Subjects Randomized | 245 | none |
| Subjects Withdrawn | 5 | none |
| Subjects who Completed the Study | 240 | none |
| Subjects Excluded from Analysis | 1 | Give Reasons |

Table 2: Number of completed pairs of injection per Comparator PN (Example only)

| Comparator | N.pairs |
|--------------------|---------|
| Artsana 33G | 265 |
| Artsana 34G | 265 |
| Simple Diagnostics | 265 |

#### 8.1.2 Data Exclusions

All exclusions will be listed with reason(s) for exclusion.

DBC-18PENDL02 



#### 8.1.3 Executive Summary

A high level summary will be provided for each objective/endpoint (example below).

# Primary Objective (examples only):

• *Injection Pain:* The lower bound of the CI for the average relative pain comparison between BD Nano<sup>™</sup> PRO and Artsana Insupen<sup>®</sup> 33G met both non-inferiority and superiority criteria.

# Secondary Objectives (examples only):

- *Injection force*: The lower bound of the CI for the average difference in rating of BD Nano<sup>™</sup> PRO and Artsana Insupen<sup>®</sup> 33G injection force met the superiority criterion.
- Needle Bending: The upper bound of the CI for the average difference in percentage of needle bending occurrence with BD Nano<sup>™</sup> PRO and Artsana Insupen<sup>®</sup> 33G met the superiority criterion.
- Leakage: The upper bound of the CI for the average difference in percentage of leakage occurrence with BD Nano™ PRO and Artsana Insupen® 33G met the superiority criterion.

In addition, a summary table for all primary and secondary objectives will be presented as in Table 3 (Example only). A blue check mark  $(\checkmark)$  indicates that the acceptance criterion is met, while a red X mark (×) indicates that the acceptance criterion is not met.

Table 3: Results Summary of primary and secondary objectives (Example only)

| Objective | Comparison | |
|----------------------------------|-------------------------------|----------|
| Primary Objective | | |
| Injection Pain (Non-inferiority) | BD Nano vs Artsana 33G | <b>✓</b> |
| Injection Pain (Non-inferiority) | BD Nano vs Artsana 34G | <b>✓</b> |
| Injection Pain (Non-inferiority) | BD Nano vs Simple Diagnostics | <b>✓</b> |
| Secondary Objective | | |
| Injection Pain (Superiority) | BD Nano vs Artsana 33G | × |
| Injection Pain (Superiority) | BD Nano vs Artsana 34G | × |
| Injection Pain (Superiority) | BD Nano vs Simple Diagnostics | × |
| Injection force | BD Nano vs Artsana 33G | <b>✓</b> |
| Injection force | BD Nano vs Artsana 34G | <b>✓</b> |
| Injection force | BD Nano vs Simple Diagnostics | <b>✓</b> |
| Needle Bending | BD Nano vs Artsana 33G | <b>✓</b> |
| Needle Bending | BD Nano vs Artsana 34G | <b>✓</b> |
| Needle Bending | BD Nano vs Simple Diagnostics | <b>✓</b> |
| Leakage | BD Nano vs Artsana 33G | ✓ |
| Leakage | BD Nano vs Artsana 34G | ✓ |
| Leakage | BD Nano vs Simple Diagnostics | <b>✓</b> |

DBC-18PENDL02 



# 8.2 Analysis and Results

# 8.2.1 Injection Pain

Summary statistics for the VAS scale will be presented as in Table 4.

The results for average relative VAS Score for BD Nano<sup> $\top$ M</sup> PRO vs comparator pen needle will be evaluated as presented in Table 5.

Table 4: Summary Statistics for observed 150mm Relative VAS Scores (Example only)

| Comparison | N | Mean | Std. Dev. | Mean 95% CI | Median | Median 95% CI | Range |
|---|---|---|---|---|---|---|---|
| BD Nano vs Artsana 33G | 13 | 12.12 | 44.00 | (-74.13, 98.36) | 15.00 | (-71.25, 101.25) | -75, 67.5 |
| BD Nano vs Artsana 34G | 12 | 0.00 | 27.14 | (-53.19, 53.19) | -7.50 | (-60.69, 45.69) | -37.5, 45 |
| BD Nano vs Simple Diagnostics | 9 | -10.00 | 41.59 | (-91.52, 71.52) | -22.50 | (-104.02, 59.02) | -52.5, 60 |

Table 5: Fitted Average Relative VAS score for BD Nano vs comparator pen needles (Example only)

| Comparison | Fitted Mean | CI | Non-Inferiority<br>Conclusion (Lower<br>bound CI > -10) | Superiority Conclusion (Lower bound $CI > 0$ ) |
|---|---|---|---|---|
| BD Nano vs Artsana 33G | 28.3 | (17.1, 39.4) | TRUE | TRUE |
| BD Nano vs Artsana 34G | 19.2 | (4.1, 34.4) | $\operatorname{TRUE}$ | TRUE |
| BD Nano vs Simple Diagnostics | 26.1 | (10.3, 42) | TRUE | TRUE |

DBC-18PENDL02 





Figure 2: Distribution of relative VAS scores with average and confidence interval per pen needle group and overall. Positive scores indicate that BD Next was preferred and negative scores indicate that the Current/Assigned PN was preferred. Note: This example graph comes from a study with different PN. Results for this study will reflect BD Nano performance.

DBC-18PENDL02 



# 8.2.2 Injection force

The distribution of the ratings of injection force for BD Nano vs each comparator pen needle will be presented as in Table 6 and Figure 3. Summary statistics for the ratings of injection force will be presented as in Table 7.

The results of average ratings will be evaluated as presented in Table 8.

Table 6: Distribution of injection force ratings (BD Nano vs Artsana 33G) (Example only)

| Rating | n (%) |
|-------------------------------------------------|-------------|
| -2 (Artsana 33G significantly less thumb force) | 66 (20.0%) |
| -1 (Artsana 33G slightly less thumb force) | 66 (20.0%) |
| 0 (No Difference) | 66 (20.0%) |
| 1 (BD Nano slightly less thumb force) | 66 (20.0%) |
| 2 (BD Nano significantly less thumb force) | 66 (20.0%) |
| Total | 330 |
| All Rating: >0 | 132 (43.9%) |

Table 7: Summary Statistics for observed ratings of injection force (Example only)

| Comparison | N | Mean | Std. Dev. | Mean 95% CI | Median | Median 95% CI | Range |
|---|---|---|---|---|---|---|---|
| BD Nano vs Artsana 33G | 266 | 1.4 | 0.1 | [-0.1, 2] | 1.5 | [-0.1, 2] | -2, 2 |
| BD Nano vs Artsana 34G | 266 | 1.5 | 0.1 | [-0.1, 2] | 1.5 | [-0.1, 2] | -2, 2 |
| BD Nano vs Simple Diagnostics | 266 | 1.6 | 0.1 | [-0.1, 2] | 1.5 | [-0.1, 2] | -2, 2 |

DBC-18PENDL02 



### Observed ratings of injection force



Figure 3: Summary for observed ratings of injection force per pen needle type (Example only)

DBC-18PENDL02 



Table 8: Fitted average ratings of injection force (Example only)

| Comparison | Mean | CI | Superiority Conclusion (Lower bound $CI > 0$ ) |
|---|---|---|---|
| BD Nano vs Artsana 33G | 1.30 | [-0.1, 2] | Fail |
| BD Nano vs Artsana 34G | 1.40 | [0.1, 2.5] | Pass |
| BD Nano vs Simple Diagnostics | 1.60 | [0.1, 2.8] | Pass |

The difference in percentage of responses with a preference for BD vs each comparator pen needle will be presented as in Table 9.

Table 9: Difference in Percentage of responses with a preference for BD Nano vs comparator PN (Example only)

| \ 1 0/ | | | | |
|---|---|---|---|---|
| Comparison | percentage of re- | percentage of re- | Difference in Percent- | 95% CI for Difference |
| | sponses with a prefer- | sponses with a prefer- | age (BD Nano - com- | |
| | ence for BD Nano | ence for comparator | parator) | |
| BD Nano vs Artsana 33G | 45.5% | 40.0% | 5.5% | [2.1%, 6.8%] |
| BD Nano vs Artsana 34G | 55.5% | 30.0% | 25.5% | [12.2%, 36.8%] |
| BD Nano vs Simple Diagnostics | 49.5% | 35.0% | 14.5% | [10.1%, 18.8%] |

#### 8.2.3 Needle Bending

Summary statistics for needle bending will be presented as in Table 10.

The results of difference in percentage of needle bending will be evaluated as presented in Table 11.

Table 10: Observed percentage of Needle Bending (Example only)

| • | O | 0 ( |
|--------------------|-------------------|--------------|
| Pen Needle | Needle bending | 95% CI |
| BD Nano | $2/266 \ (0.8\%)$ | [0.1%, 1.5%] |
| Artsana 33G | $5/266 \ (1.9\%)$ | [1.2%, 2.6%] |
| Artsana 34G | 5/266~(1.9%) | [1.2%, 2.6%] |
| Simple Diagnostics | $5/266 \ (1.9\%)$ | [1.2%, 2.6%] |

Table 11: Difference in Percentage of Needle Bending based on modeling analysis. (Example only)

| Comparison | Difference in Percentage of Needle bending | 95% CI for Difference | Superiority (Upper bound <0) |
|---|---|---|---|
| BD Nano vs Artsana 33G | -1.1% | [-3.2%, 0.8%] | Fail |
| BD Nano vs Artsana 34G | -1.1% | [-3.2%, 0.8%] | Fail |
| BD Nano vs Simple Diagnostics | -1.1% | [-3.2%, 0.8%] | Fail |

#### 8.2.4 Leakage from Injection Site

Summary statistics for leakage from injection site will be presented as in Table 12. The distribution of leakage from injection site will be presented as in Figure 4.

The leakage on a binary scale will also be presented and analyzed as in Section 8.2.3.

DBC-18PENDL02 



Table 12: Summary Statistics for leakage from injection site (Example only)

| Pen needle | N | Mean | Std. Dev. | Median | Range |
|--------------------|---|--------|-----------|--------|-----------------|
| BD Nano | 3 | 0.0176 | 0.0189 | 0.0185 | 0.0112,0.0298 |
| Artsana 33G | 5 | 0.0234 | 0.0147 | 0.0226 | 0.0132,0.0342 |
| Artsana 34G | 6 | 0.0234 | 0.0147 | 0.0226 | 0.0132, 0.0342 |
| Simple Diagnostics | 6 | 0.0234 | 0.0147 | 0.0226 | 0.0132,0.0342 |



Figure 4: Leakage from the injections per pen needle type. The blue line represents the threshold for leakage (0.015g).

DBC-18PENDL02 



# 8.2.5 Exploratory Objectives

Patient end needle breaking will be summarized as in Section 8.2.3.

Summary statistics for delivery time and total injection time will be presented as in Table 13. The average difference (BD PN - comparator PN) in delivery time and total injection time will be evaluated as presented in Table 14.

Summary statistics for Non-Comparative Questionnaire will be presented as in Table 7.

Table 13: Summary Statistics for delivery time (Example only)

| Pen Needle | N | SD | Mean | Median | Range |
|--------------------|----|-------|--------|--------|----------|
| BD Nano | 31 | 40.52 | 142.03 | 142.00 | 90, 274 |
| Artsana 33G | 31 | 63.90 | 165.84 | 140.00 | 91, 362 |
| Artsana 34G | 29 | 46.64 | 150.41 | 137.00 | 84, 324 |
| Simple Diagnostics | 30 | 56.14 | 171.20 | 150.00 | 103, 322 |

Table 14: Mean difference of Delivery time and Total injection time with confidence interval (reciprocal of number of seconds) between BD Nano and Artsana 33G. The last column indicates whether superiority was met or not. (Example only)

| | Mean difference | 95% Lower bound | P value | Superiority (Lower bound >0) |
|---|---|---|---|---|
| Delivery time | -0.000739 | -0.001658 | 0.113 | Fail |
| Total injection time | 0.000452 | -0.000377 | 0.279 | Fail |

# 8.3 Demographics and Diabetes History

Table 15: Subject Demographics (Example only)

| | <b>J</b> | , 1 | ( | |
|------|---------------|-------|------------------|--------------------------|
| Char | acteristic | | Resul | $\overline{\mathrm{ts}}$ |
| Gend | er | | | |
| | Female | | 94 (50 | 0.8% |
| | Male | | 91 (49 | 9.2% |
| Age | | | ` | , |
| | Mean | | 55.8 | |
| | 95% Mean CI | | 53.9, | 57.7 |
| | SD | | $13.0^{\circ}$ | |
| | Min, Max | | 20, 76 | ; |
| | Observation ( | Count | $18\overline{3}$ | |
| | Missing Coun | t | 2 | |
| | Total Count | | 185 | |

Table 16: Distribution of Type of Diabetes (Example only)

| Characteristic | Results |
|---|---|
| Diabetes Type<br>Type II<br>Type I<br>Missing | 152 (84.4%)<br>28 (15.6%)<br>2 |

DBC-18PENDL02 



Table 17: Diabetes History (Example only)

| Table 11. Diabetes History (Examp | ne omy |
|-----------------------------------|----------------|
| Characteristic | Results |
| Diagnosed year | |
| Mean | 14.2 |
| 95% Mean CI | 12.8, 15.6 |
| $\operatorname{SD}$ | 9.4 |
| Min, Max | 1, 54 |
| Total Count | 182 |
| Injection Times per day | |
| once | 74 (40.7%) |
| four | 36 (19.8%) |
| twice | $31\ (17.0\%)$ |
| five or more | 19 (10.4%) |
| NA - injects non-insulin only | 11 ( 6.0%) |
| three | 11 ( 6.0%) |
| Pen needle used | |
| BD Nano 32Gx4mm | 66 (36.5%) |
| NovoFine 32Gx6mm | 33 (18.2%) |
| Other 32G | 24 (13.3%) |
| Other 31Gx5mm | 22(12.2%) |
| NovoTwist 32Gx5mm | 20 (11.0%) |
| NovoFine Plus 32Gx4mm | 14 ( 7.7%) |
| Owen Mumford PenTips 32Gx4mm | 2 (1.1%) |
| Missing | 1 |
| Injection site used | |
| Abdomen | 158 (87.3%) |
| Thigh | 14 ( 7.7%) |
| Arm | 7 (3.9%) |
| Buttocks | 1 (0.6%) |
| Other | 1(0.6%) |
| Missing | 1 |

DBC-18PENDL02 



# 9 Appendix

# 9.1 Discontinued Data

The Table 18 shows the detailed list of discontinued subjects.

Table 18: Details of Discontinued Subjects (Example only)

| Subject ID | Completion Date | Discontinuation Time | Reason for Discontinuation | Details |
|---|---|---|---|---|
| R003 | January 3, 2018 | After initiation of study | Other | Subject decided not con- |
| | | procedure/ intervention | | tinue to participate |
| R067 | February 7, 2018 | Before any study proce- | Did not meet criteria | |
| | | dure/ intervention | (Screen Failure) | |
| R114 | February 19, 2018 | After initiation of study | Administrative Issue | Detail of reason for discon- |
| | | procedure/ intervention | | tinuation |

# 9.2 Missing Data

All the Missing data will be listed.

### 9.3 Adverse Events

Data listings will be provided for any adverse events and serious adverse event in Table 19. Adverse events will be summarized descriptively by pen needle in Table 20 and 21.

Table 19: Data listing for adverse events (Example only)

| Random | PN Used | Seriousness | Severity | Relation to | Contribution | Relation to | Description |
|---|---|---|---|---|---|---|---|
| ID | | | | product | of product | protocol | |
| | | | | | malfunction | | |
| R055 | BD Nano | Serious | Moderate | Related | Yes | Not related | adverse event to be described |
| R001 | Artsana | Serious | Mild | Unlikely re- | No | Possibly re- | adverse event to be described |
| | 33G | | | lated | | lated | |
| R099 | Artsana | Serious | Severe | Possibly re- | Yes | related | adverse event to be described |
| | 33G | | | lated | | | |

Table 20: Summary of Adverse Events: Relationship to product (Example only)

| | v | | | | ` 1 | . , |
|---|---|---|---|---|---|---|
| Pen Needle | Number of | Number of | Not related | Unlikely re- | Possibly re- | Related |
| | events | Subjects | | lated | lated | |
| BD Nano | 5 | 2 | 2 | 1 | 1 | 1 |
| Artsana 33G | 0 | 0 | 0 | 0 | 0 | 0 |
| Artsana 34G | 0 | 0 | 0 | 0 | 0 | 0 |
| Simple Diagnostics | 0 | 0 | 0 | 0 | 0 | 0 |

DBC-18PENDL02 



Table 21: Summary of Adverse Events: Relationship to protocol / procedure (Example only)

| Pen Needle | Number of | Number of | Not related | Unlikely re- | Possibly re- | Related |
|---|---|---|---|---|---|---|
| | events | Subjects | | lated | lated | |
| BD Nano | 5 | 2 | 2 | 1 | 1 | 1 |
| Artsana 33G | 0 | 0 | 0 | 0 | 0 | 0 |
| Artsana 34G | 0 | 0 | 0 | 0 | 0 | 0 |
| Simple Diagnostics | 3 | 3 | 0 | 1 | 0 | 2 |

DBC-18PENDL02 